CLINICAL TRIAL: NCT05642494
Title: Comparison of the Effectiveness of Silver Diamine Fluoride Versus Silver Diamine Fluoride Combined With Sodium Fluoride Varnish in the Arrest of Early Childhood Caries: A Randomised Controlled Clinical Trial
Brief Title: Silver Diamine Fluoride(SDF) Versus SDF Combined With Sodium Fluoride Varnish in the Arrest of Early Childhood Caries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Science, Technology & Innovation Funding Authority (STDF) (Unknown)
Responsible Party: Principal Investigator, Enas Belal, Instructor of Dental Public Health, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0272-07/2021
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Early Childhood Caries
Keywords: ECC; SDF 38%; NaF 5%; preschoolers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SDF+NaF (Experimental): Silver Diamine fluoride 38% (Applied biannually)+ Sodium Fluoride Varnish 5% (Applied every 3 months)
  Interventions: Device: SDF; Device: NaF
- SDF (Active Comparator): Silver Diamine fluoride 38% (Applied biannually)
  Interventions: Device: SDF

INTERVENTIONS:
Device: SDF — Silver Diamine Fluoride 38% (Applied bianually)
Device: NaF — Sodium Fluoride Varnish (5%) (Applied at baseline and after 3 months)
  Arms: SDF+NaF

SUMMARY:
Early childhood caries (ECC) is the most common chronic childhood disease worldwide. Early restorative intervention may treat the disease but this is often difficult especially with uncooperative children so it may be left untreated. Remineralization of affected dentin using silver diamine fluoride (SDF) can arrest these lesions.

This trial aims to compare the effectiveness of 38% SDF solution versus 38% SDF solution with 5% sodium fluoride (NaF) varnish after six months in arresting ECC lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Children ≤ 4 years old.
2. The presence of at least one carious lesion on a primary tooth, with scores 3 and higher (according to the International Detection and Assessment System- ICDAS II, Appendix 1, Table 1), detected by visual examination.
3. The Carious lesion has to be active according to Lesion Activity criteria of coronal caries of ICDAS II.
4. Parental consent for children's participation in the study.

Exclusion Criteria:

1. Children reporting spontaneous or elicited pain from caries, or showing any signs of pulpal infection, swelling and/or abscess.
2. Children showing a definite negative behavior (Score 1 Frankel's classification) during clinical examination.
3. Allergy or sensitivity to silver or any of the materials included in the study.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The percentage of arrested carious lesions | 6 months
  For cavitated dentine caries lesions diagnosed as ICDAS code 5 or 6, visual inspection and tactile detection using a 0.5mm ball-ended Community Periodontal Index (CPI) probe without radiograph examination will be used for assessing caries activity according to Lesion Activity criteria of ICDAS II. If a wall or floor of the lesion is soft and easily penetrated by the probe using light force, then it will be diagnosed as active. A lesion with all surfaces being hard and smooth will be diagnosed as arrested caries .For a moderate caries lesion with no visible dentine (ICDAS code 3 or 4) at baseline, it will be classified as arrested caries at follow-up examination if the lesion did not progress to become a cavitated lesion with visible dentine (ICDAS code 5 or 6). Five tooth surfaces (buccal, lingual, mesial, distal and occlusal) will be examined in each posterior tooth and 4 tooth surfaces (labial, lingual, mesial and distal) in each anterior tooth.

SECONDARY OUTCOMES:
Caries Increment (number of new caries lesions) | 6 months
  New caries lesions will be assessed through visual and tactile inspection using the World Health Organization (WHO) criteria for caries diagnosis. Full mouth examination will be conducted with the aid of a WHO CPI probe, and a disposable dental mirror. Five tooth surfaces (buccal, lingual, mesial, distal and occlusal) will be examined in each posterior tooth and 4 tooth surfaces (labial, lingual, mesial and distal) in each anterior tooth to assess the caries increment using the decayed, missing (due to caries), and filled primary tooth index per surface (dmfs).
Parental satisfaction with SDF application | Baseline and at 6 months
  Parents will be asked If SDF Application is an easy process. Answers will be on a 5 point Likert scale (Strongly agree, Agree Neutral , Disagree, Strongly disagree).
Parental satisfaction with SDF application | Baseline and at 6 months
  Parents will be asked if they are comfortable with discoloration of cavities after SDF placement, Answers will be on a 5 point Likert scale (Strongly agree, Agree Neutral , Disagree, Strongly disagree).
Parental satisfaction with SDF application | Baseline and at 6 months
  Parents will be asked If SDF application was pain free for their child .Answers will be on a 5 point Likert scale (Strongly agree, Agree Neutral , Disagree, Strongly disagree).
Parental satisfaction with SDF application | Baseline and at 6 months
  Parents will be asked if The taste of SDF was acceptable to their child.Answers will be on a 5 point Likert scale (Strongly agree, Agree Neutral , Disagree, Strongly disagree).
Adverse effects reported after application of the interventions | Baseline and at 6 months
  Parents will be asked if their child experienced tooth or gum pain after application of the material.
  (Yes/No) Question
Adverse effects reported after application of the interventions | Baseline and at 6 months
  The clinician will observe if gum swelling occurred after application of the material.
  (Yes/No) Question
Adverse effects reported after application of the interventions | Baseline and at 6 months
  The clinician will observe if gum bleaching occurred after application of the material.
  (Yes/No) Question
Adverse effects reported after application of the interventions | Baseline and at 6 months
  Systemic toxicity (nausea, vomiting, generalised discomfort) will be assesses by the clinician at the time of application and by asking the parents one week later.
  (Yes/No) Question
Adverse effects reported after application of the interventions | Baseline and at 6 months
  Black staining of each lesion will be clinically observed and recorded (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Enas B Abdellatif, Bachelor, Principal Investigator — Alexandria University
Locations (1):
- Faculty Of Dentistry Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdellatif EB, El Kashlan MK, El Tantawi M. Silver diamine fluoride with sodium fluoride varnish versus silver diamine fluoride in arresting early childhood caries: a 6-months follow up of a randomized field trial. BMC Oral Health. 2023 Nov 17;23(1):875. doi: 10.1186/s12903-023-03597-5. PMID 37978488